CLINICAL TRIAL: NCT07252414
Title: A Phase 1, Multicenter, Open-Label, First-in-Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-Tumor Activity of GenSci143 in Participants With Advanced Solid Tumors
Brief Title: GenSci143 in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GenSci143-101
Record Dates: First submitted 2025-11-14; First posted 2025-11-26 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GenSci143 for injection (Experimental)
  Interventions: Drug: GenSci143 for injection

INTERVENTIONS:
Drug: GenSci143 for injection — GenSci143 for injection, administered Q3W, with a dosage ranging from 0.5mg/kg to 4.5mg/kg.

SUMMARY:
A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-Tumor Activity of GenSci143 in Participants with Advanced Solid Tumors

DETAILED DESCRIPTION:
A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-Tumor Activity of GenSci143 in Participants with Advanced Solid Tumors

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign the ICF.
* Male or female participants ≥18 years old at the time of signing the ICF.
* Meet the requirements of tumor types as outlined below:

  1. Dose escalation: Participants with histologically or cytologically documented recurrent or metastatic advanced solid tumors, and who have progressed after standard therapy, are intolerant to standard therapy, or have no standard therapy available.
  2. Dose expansion:

Cohort 1: Participants with histologically or cytologically documented mCRPC，who had received at least one prior novel hormonal therapy (including but not limited to abiraterone, enzalutamide, darolutamide, apalutamide) and progressed on standard chemotherapy regimens, are intolerant to chemotherapy, or decline chemotherapy.

Cohort 2: Participants with histologically or cytologically documented other advanced solid tumors, and who have progressed after standard therapy, are intolerant to standard treatment, or have no standard therapy available.

* Life expectancy of ≥ 12 weeks.
* ECOG PS 0-1
* Have at least 1 evaluable tumor lesion according to RECIST v1.1. Participants with mCRPC who have bone only disease may be eligible on a case-by-case basis after discussion between the investigator and Sponsor
* Able to provide either archival or fresh biopsy formalin-fixed paraffin-embedded (FFPE) tumor samples.
* Adequate organ function at the time of screening, as outlined below:

  1. Hematology: Absolute neutrophil count (ANC) ≥ 1.5×109/L (1500/µL); platelet count (PLT)≥100×109/L (100,000/µL); hemoglobin (HGB) ≥ 90 g/L (9 g/dL) (have not received granulocyte colony-stimulating factor (G-CSF) within 7 days before the first dose of GenSci143, and have not received granulocyte-macrophage colony-stimulating factor (GM-CSF), blood transfusion, erythropoietin (EPO), platelet transfusion, thrombopoietin (TPO), or interleukin-11 (IL-11) within 14 days before the first dose of GenSci143).
  2. Liver function: Serum total bilirubin (TBIL) ≤ 1.5 upper limit of normal (ULN), and serum TBIL≤ 3×ULN in the presence of liver metastasis or documented Gilbert syndrome. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3×ULN if no liver metastasis; ALT and AST≤ 5×ULN in the presence of liver metastasis.
  3. Renal function: creatinine clearance (CLcr) ≥ 50 mL/min as calculated using the Cockcroft-Gault formula.
  4. Coagulation function: Prothrombin Time (PT), activated partial thromboplastin time (APTT), and international normalized ratio (INR) ≤ 1.5×ULN (or within target range if on anticoagulation therapy).
* Toxicities (other than alopecia) from previous anticancer therapy must have resolved to NCI-CTCAE v5.0 Grade ≤1.
* Women of childbearing potential (WOCBP) must have a serum pregnancy test negative within 7 days before the first dose of GenSci143. WOCBP must agree to use highly effective contraceptive methods and must not donate or retrieve ova for personal use from the time of informed consent until 6 months after the last dose of GenSci143. Male participants must agree to use highly effective contraceptive methods and must not freeze or donate sperm from the time of informed consent until 6 months after the last dose of GenSci143.

Exclusion Criteria:

* Participants with known spinal cord compression or active central nervous system (CNS) metastases, unless they are asymptomatic or have achieved post-treatment stability for >4 weeks and discontinued corticosteroids for >2 weeks before the first dose of GenSci143.
* History of other known malignancies within the past 3 years.
* Unstable thrombotic events requiring therapeutic intervention within 6 months before the first dose of GenSci143.
* Uncontrolled or clinically significant cardiovascular disease.
* Uncontrolled pleural fluid, pericardial effusion, or ascites requiring drainage, and/or diuretics within 2 weeks before the first dose of GenSci143.
* History of (non-infectious) interstitial lung disease (ILD)/pneumonitis that requires steroids, current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at Screening. Any autoimmune, connective tissue, or inflammatory disorders with suspected pulmonary involvement.
* Pregnant, breastfeeding, or planning to become pregnant.
* Known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
* Known human immunodeficiency virus (HIV) infection
* Uncontrolled infection that requires systemic therapy with IV antibiotics, antivirals, or antifungals within 1 week before the first dose of GenSci143.
* Major surgery (excluding diagnostic surgery), radiotherapy, and immunotherapy within 4 weeks before the first dose of medication; Chemotherapy or antibody therapy within 3 weeks; Endocrine therapy and small molecule-targeted therapy within 2 weeks or 5 half-lives(whichever is shorter). Androgen-deprivation therapy with gonadotropin-releasing hormone (GnRH) analogues (either GnRH agonists or GnRH antagonists) was allowed for men with prostate cancer.
* Received any live vaccine within 4 weeks before the first dose of GenSci143 or intend to receive a live vaccine during the study.
* History of allogeneic hematopoietic stem cell transplantation (HSCT) or solid organ transplantation.
* Prior treatment with a topoisomerase inhibitor or an ADC that consists of a topoisomerase inhibitor.
* History of severe hypersensitivity reactions to GenSci143 and/or excipients in the drug product, or other monoclonal antibodies.
* Any illness (uncontrolled hypertension, serious diabetes mellitus, thyroid disorders, and psychiatric disorders, etc.) or other conditions that are not eligible for inclusion based on the investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-12-20 (Actual); Primary Completion 2028-10-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Part 1 and Part2:Incidence of adverse events Percentage of patients with adverse events by system organ class and preferred term. | From time of informed consent to 30days post last dose of GenSci143
Part1:Dose limiting toxicities(DLTs),DLTs are assessed during the DLT observation period and defined as any toxicity in DLT definition in the Clinical Study Protocal | Form time of first dose of GenSci143 to end of DLT observation period(approximately 21 days)
Part1: Maximum tolerated dose (MTD) and recommended dose for expansion (RDE) To determine the maximum tolerated dose (MTD) (if applicable) and recommended dose for expansion (RDE) of GenSci143. | Form time of first dose of GenSci143 up to 12 months.
Part1: Part2: Composite response rate To evaluate the efficacy of GenSci143 as using RECIST v1.1 and/or PSA50 response (PCWG3) with PC | Approximately 12 months.
Part1: Part2: Objective response rate(ORR) To evaluate the efficacy of GenSci143 as measured by ORR using RECIST v1.1 for participants with non-PC | Approximately 12 months.

SECONDARY OUTCOMES:
AUC of GenSci143 Calculate area under the curve of GenSci143. | Approximately 12 months.
AUC of total antibody Calculate area under the curve of total antibody. | Approximately 12 months

OTHER OUTCOMES:
AUC of unconjugated payload. Calculate area under the curve of unconjugated payload | Approximately 12 months
Cmax of GenSci143 Calculate maximum concentration of GenSci143. | Approximately 12 months
Cmax of total antibody Calculate maximum concentration of total antibody | Approximately 12 months
Cmax of unconjugated payload Calculate maximum concentration of unconjugated payload | Approximately 12 months
Tmax of GenSci143 Calculate time of maximum concentration of GenSci143 | Approximately 12 months
Tmax of total antibody Calculate time of maximum concentration of total antibody | Approximately 12 months
Tmax of unconjugated payload Calculate time of maximum concentration of unconjugated payload | Approximately 12 months
CL of GenSci143 Calculate Cleanrance of GenSci143 | Approximately 12 months
CL of total antibody Calculate Cleanrance of total antibody | Approximately 12 months
CL of unconjugated payload Calculate Cleanrance of unconjugated payload | Approximately 12 months
V of GenSci143 Calculate apparent volume of distribution of GenSci143 | Approximately 12 months
V of total antibody Calculate apparent volume of distribution of total antibody | Approximately 12 months
V of unconjugated payload Calculate apparent volume of distribution of unconjugated payload | Approximately 12 months
t1/2 of GenSci143 Calculate time of half-life of GenSci143 | Approximately 12 months
t1/2 of total antibody Calculate time of half-life of total antibody | Approximately 12 months
t1/2 of unconjugated payload Calculate time of half-life of unconjugated payload | Approximately 12 months
ADC of GenSci143 Incidence and titer of anti-drug antibody(ADA) | Approximately 12 months
NAb of GenSci143 Incidence and titer of anti-drug neutralizing(NAb) | Approximately 12 months
Prostate-specific antigen (PSA)50 response rate To evaluate the preliminary anti-tumor activity of GenSci143 by PSA50 as PCWG3 criteria and RECIST v1.1 with PC | Approximately 12 months
PSA90 response rate To evaluate the preliminary anti-tumor activity of GenSci143 by PSA90 as PCWG3 criteria and RECIST v1.1 with PC. | Approximately 12 months
Best PSA response To evaluate the preliminary anti-tumor activity of GenSci143 by best PSA response as PCWG3 criteria and RECIST v1.1 with PC. | Approximately 12 months
PSA progression-free survival (PSA-PFS) To evaluate the preliminary anti-tumor activity of GenSci143 by PSA-PFS as PCWG3 criteria and RECIST v1.1 with PC. | Approximately 12 months
radiological PFS (rPFS) To evaluate the preliminary anti-tumor activity of GenSci143 by rPFS as PCWG3 criteria and RECIST v1.1 with PC. | Approximately 12 months
failure-free survival (FFS) To evaluate the preliminary anti-tumor activity of GenSci143 by FFS as PCWG3 criteria and RECIST v1.1 with PC. | Approximately 12 months
overall survival (OS) To evaluate the preliminary anti-tumor activity of GenSci143 by OS as PCWG3 criteria and RECIST v1.1 with PC. | Approximately 12 months
objective response rate (ORR) To evaluate the preliminary anti-tumor activity of GenSci143 by ORR as PCWG3 criteria and RECIST v1.1 with PC. | Approximately 12 months
disease control rate (DCR) To evaluate the preliminary anti-tumor activity of GenSci143 by DCR as PCWG3 criteria and RECIST v1.1 with PC. | Approximately 12 months
duration of response (DoR) To evaluate the preliminary anti-tumor activity of GenSci143 by DoR as PCWG3 criteria and RECIST v1.1 with PC. | Approximately 12 months
time to response (TTR) To evaluate the preliminary anti-tumor activity of GenSci143 by TTR as PCWG3 criteria and RECIST v1.1 with PC. | Approximately 12 months
depth of response (DpR) To evaluate the preliminary anti-tumor activity of GenSci143 by DpR as PCWG3 criteria and RECIST v1.1 with PC. | Approximately 12 months
overall survival (OS) To evaluate the preliminary anti-tumor activity of GenSci143 by OS as RECIST v1.1 with non-PC. | Approximately 12 months
objective response rate (ORR) To evaluate the preliminary anti-tumor activity of GenSci143 by ORR as RECIST v1.1 with non-PC. | Approximately 12 months
disease control rate (DCR) To evaluate the preliminary anti-tumor activity of GenSci143 by DCR as RECIST v1.1 with non-PC. | Approximately 12 months
duration of response (DoR) To evaluate the preliminary anti-tumor activity of GenSci143 by DoR as RECIST v1.1 with non-PC. | Approximately 12 months
time to response (TTR) To evaluate the preliminary anti-tumor activity of GenSci143 by TTR as RECIST v1.1 with non-PC. | Approximately 12 months
depth of response (DpR) To evaluate the preliminary anti-tumor activity of GenSci143 by DpR as RECIST v1.1 with non-PC. | Approximately 12 months

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Shandong Cancer Hospital, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided